CLINICAL TRIAL: NCT03139136
Title: A 12-Week, Double-Blind, Placebo-Controlled, Phase 2a Study to Investigate the Safety, Tolerability and Efficacy of MBS2320 in Patients With Active Rheumatoid Arthritis Receiving Methotrexate
Brief Title: Safety, Tolerability and Efficacy of MBS2320 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Modern Biosciences Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 120012A; 2016-004038-24 (EudraCT Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBS2320 (Active Comparator)
  Interventions: Drug: MBS2320
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBS2320 — As described in the arm descriptions
  Arms: MBS2320
Drug: Placebo — As described in the arm descriptions
  Arms: Placebo

SUMMARY:
Rheumatoid arthritis (RA) affects 1 percent of the population worldwide and up to 40 percent of patients don't respond to current treatments. MBS2320, the drug being tested in this trial, represents a new approach to treating RA, with the potential not only to reduce levels of inflammation but to also directly prevent bone damage.The aim of this project is to test the safety, tolerability and efficacy of MBS2320 in patients with RA in combination with an existing treatment, methotrexate.

DETAILED DESCRIPTION:
Rheumatoid Arthritis is a chronic autoimmune disease characterised by synovial inflammation and cartilage and bone degradation, leading to joint destruction and progressive disability.

The aim of the study is to evaluate the safety and tolerability of MBS2320 in patients with RA following chronic administration. In addition, the study aims to evaluate the effects of MBS2320 on measures of disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of childbearing or non-childbearing potential with with active RA, receiving stable once-weekly methotrexate
* between 18 and 75 years of age, inclusive.

Exclusion Criteria:

* Patients who are currently pregnant or breastfeeding.
* Patients who are being treated with biological or non-biological disease-modifying anti-rheumatic drug therapy.
* Patients with a history of any other inflammatory or arthritic disease in addition to RA that may interfere with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | 12 weeks
  Incidence of all grade adverse events

SECONDARY OUTCOMES:
Disease Activity Score 28 (DAS28) | 12 weeks
  Disease Activity Score according to the EULAR response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Inga Bodrug, MD, Principal Investigator — Arensia Exploratory Medicine
Locations (3):
- Arensia, Tbilisi, Georgia
- Arensia, Chisinau, Moldova
- Arensia, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No